CLINICAL TRIAL: NCT01187329
Title: The Effect of the Hyperinsulinemic Normoglycemic Clamp on Myocardial Function and Utilization of Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-526
Record Dates: First submitted 2010-08-19; First posted 2010-08-24 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-10

CONDITIONS: Hyperglycemia; Aortic Valve Replacement; Aortic Stenosis; Cardiac Surgery
Keywords: Hyperglycemia; open heart surgery; bypass
MeSH Terms: conditions — Hyperglycemia; Aortic Valve Stenosis | interventions — Control Groups; Glucose; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hyperinsulinemic normoglycemic clamp (HNC) (Experimental): Patients will be randomized to receive treatment with HNC during cardiac surgery.
  Interventions: Other: hyperinsulinemic normoglycemic clamp (HNC)
- standard glucose management (Placebo Comparator): Patients will be randomized to receive treatment with standard glucose management during cardiac surgery.
  Interventions: Other: control group

INTERVENTIONS:
Other: hyperinsulinemic normoglycemic clamp (HNC) — Prior to anesthetic induction, a baseline blood glucose value will be obtained, followed by an insulin infusion of 5 mU.Kg-1.min-1. When blood glucose is <110 mg/dL, a variable continuous infusion of glucose (dextrose 20%) supplemented with potassium (40 mEq/L) and phosphate (30 mmol/L) is administered to preserve normoglycemia (80-110 mg/dL). The glucose infusion is titrated to target glucose levels by checking blood glucose every 5 - 15 min with Accu-Check (Roche Diagnostics, Switzerland) glucose monitor. At sternal closure, insulin infusion is decreased to 1 mU/Kg/min. On admission to the ICU, insulin treatment follows the ICU protocol. The dextrose infusion is slowly weaned off over 2 - 4 hrs maintaining blood glucose > 80 mg/dL. Arterial blood glucose is measured every 30 - 60 min for 2 hrs, then, as stated in ICU protocol.
  Arms: hyperinsulinemic normoglycemic clamp (HNC)
Other: control group — Baseline arterial blood glucose will be obtained before anesthetic induction. Repeat measurements are performed every 30-90 min. Glucose >150 on CPB will receive insulin according to intraoperative protocol. After surgery, insulin is given according to ICU protocol. Target glucose < 180 mg/dL.
  Other Names: glucose; standard of care
  Arms: standard glucose management

SUMMARY:
The overall research plan is to test the hypothesis that intraoperative treatment of hyperinsulinemic normoglycemic clamp (HNC) in cardiac surgical patients improves myocardial function and short-term outcomes compared with standard glucose management.

DETAILED DESCRIPTION:
Specific Aim #1:To determine whether intraoperative use of HNC affords cardioprotective benefits measured by improved echocardiographic measures of myocardial function, serum markers of cardiomyocyte injury, and hemodynamic indices measured immediately (at end of surgery) and during the short-term (initial hospitalization).

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 84 years old, Aortic stenosis, Scheduled for Aortic valve replacement.

Exclusion Criteria:

* Poor quality echocardiographic images unsuitable for analysis
* Off -pump surgical procedure
* Anticipated deep hypothermic circulatory arrest
* Any contraindications to transesophageal echocardiogram (TEE) or other proposed intervention
* Unable to give written informed consent (non-English speaking, vulnerable patients, etc.)

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andra Duncan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Zhang K, Kumar N, Alfirevic A, Sale S, You J, Bauer A, Duncan AE. Left Ventricular Twist Mechanics Before and After Aortic Valve Replacement: A Feasibility Study and Exploratory Analysis. Semin Cardiothorac Vasc Anesth. 2022 Sep;26(3):226-236. doi: 10.1177/10892532221114791. Epub 2022 Jul 18. PMID 35848424
- [Derived] Zhang K, Sheu R, Zimmerman NM, Alfirevic A, Sale S, Gillinov AM, Duncan AE. A Comparison of Global Longitudinal, Circumferential, and Radial Strain to Predict Outcomes After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 May;33(5):1315-1322. doi: 10.1053/j.jvca.2018.10.031. Epub 2018 Oct 24. PMID 30581109
- [Derived] Sonny A, Alfirevic A, Sale S, Zimmerman NM, You J, Gillinov AM, Sessler DI, Duncan AE. Reduced Left Ventricular Global Longitudinal Strain Predicts Prolonged Hospitalization: A Cohort Analysis of Patients Having Aortic Valve Replacement Surgery. Anesth Analg. 2018 May;126(5):1484-1493. doi: 10.1213/ANE.0000000000002684. PMID 29200066
- [Derived] Duncan AE, Sarwar S, Kateby Kashy B, Sonny A, Sale S, Alfirevic A, Yang D, Thomas JD, Gillinov M, Sessler DI. Early Left and Right Ventricular Response to Aortic Valve Replacement. Anesth Analg. 2017 Feb;124(2):406-418. doi: 10.1213/ANE.0000000000001108. PMID 26702865

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperinsulinemic Normoglycemic Clamp (HNC) | Standard Glucose Management
Started | 50 | 50
Completed | 49 | 48
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperinsulinemic Normoglycemic Clamp (HNC) | Standard Glucose Management | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9) | 70 (11) | 70 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 36 | 31 | 67

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Function: Left Ventricular Global Longitudinal Strain (%)
Description: Left ventricular global longitudinal strain measured by intraoperative transesophageal echocardiography at end of surgery and assessed using off-line speckle-tracking echocardiography.
  higher values (%) mean a worse outcome.
Time Frame: end of surgery (closure), an average of 5 minutes
Population: some patient's echocardiography were low quality and can not be used
Measure: Mean (Standard Deviation); unit: percentage of myocardial shortening
Arm/Group | Hyperinsulinemic Normoglycemic Clamp (HNC) | Standard Glucose Management
Number analyzed (Participants) | 36 | 36
percentage of myocardial shortening | -16.8 (4.6) | -15.9 (4.6)
Statistical Analysis 1: Comparison: Hyperinsulinemic Normoglycemic Clamp (HNC) vs Standard Glucose Management; Test type: Superiority; p = 0.11, t-test, 2 sided; Mean Difference (Final Values) = -1.2, 97.5% CI 2-sided [-2.87 to 0.48]

2. Primary Outcome: Intraoperative Left Ventricular (LV) Global Longitudinal Strain Rate
Description: Left ventricular global longitudinal strain rate measured by intraoperative transesophageal echocardiography at end of surgery and assessed using off-line speckle-tracking echocardiography.
  higher values mean a worse outcome
Time Frame: end of surgery (closure) an average of 5 minutes
Population: some patient's echocardiography were low quality and can not be used
Measure: Mean (Standard Deviation); unit: Percent / sec
Arm/Group | Hyperinsulinemic Normoglycemic Clamp (HNC) | Standard Glucose Management
Number analyzed (Participants) | 33 | 34
Percent / sec | -1.1 (0.3) | -1.0 (0.3)
Statistical Analysis 1: Comparison: Hyperinsulinemic Normoglycemic Clamp (HNC) vs Standard Glucose Management; Test type: Superiority; p = 0.007, t-test, 2 sided; paired t-test; Mean Difference (Final Values) = -0.2, 97.5% CI 2-sided [-0.3 to -0.01]

3. Secondary Outcome: Intraoperative Right Ventricular (RV) Systolic Longitudinal Strain
Description: Right ventricular global longitudinal strain measured by intraoperative transesophageal echocardiography at end of surgery and assessed using off-line speckle-tracking echocardiography.
  higher values mean a worse outcome.
Time Frame: end of surgery (closure) an average of 5 minutes
Population: some patient's echocardiography were low quality and can not be used
Measure: Mean (Standard Deviation); unit: percentage of myocardial shortening
Arm/Group | Hyperinsulinemic Normoglycemic Clamp (HNC) | Standard Glucose Management
Number analyzed (Participants) | 26 | 28
percentage of myocardial shortening | -17.2 (4.3) | -17.3 (3.7)
Statistical Analysis 1: Comparison: Hyperinsulinemic Normoglycemic Clamp (HNC) vs Standard Glucose Management; Test type: Superiority; p = 0.57, t-test, 2 sided; Median Difference (Final Values) = -0.6, 95% CI 2-sided [-2.6 to 1.5]

4. Secondary Outcome: Intraoperative Right Ventricular (RV) Systolic Longitudinal Strain Rate
Description: Right ventricular global longitudinal strain rate measured by intraoperative transesophageal echocardiography at end of surgery and assessed using off-line speckle-tracking echocardiography.
  higher values mean a worse outcome
Time Frame: end of surgery (closure) an average of 5 minutes
Population: some patient's echocardiography were low quality and can not be used
Measure: Mean (Standard Deviation); unit: Percent / sec
Arm/Group | Hyperinsulinemic Normoglycemic Clamp (HNC) | Standard Glucose Management
Number analyzed (Participants) | 26 | 28
Percent / sec | -1.1 (0.3) | -1.1 (0.4)
Statistical Analysis 1: Comparison: Hyperinsulinemic Normoglycemic Clamp (HNC) vs Standard Glucose Management; Test type: Superiority; p = 0.45, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.1]

ADVERSE EVENTS:
Arm/Group | Hyperinsulinemic Normoglycemic Clamp (HNC) | Standard Glucose Management
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 0/49 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No